CLINICAL TRIAL: NCT06459284
Title: Instrument Tissue Interaction at the Grasp Site During Membrane Peeling of Epiretinal Membranes - a Retrospective Exploratory Study
Brief Title: Instrument Tissue Interaction at the Grasp Site During Membrane Peeling of Epiretinal Membranes
Status: Completed | Type: Observational
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: ITI
Record Dates: First submitted 2024-06-02; First posted 2024-06-14 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early use of iOCT group: Patients having undergone pars plana vitrectomy with membrane Peeling die to an epiretinal Membrane in the time period from 1.6.2014 to 31.12.2016.
  Interventions: Other: retrospective data analysis
- later use of iOCT group: Patients having undergone pars plana vitrectomy with membrane Peeling die to an epiretinal Membrane in the time period from 1.11.2020 to 31.7.2022.
  Interventions: Other: retrospective data analysis

INTERVENTIONS:
Other: retrospective data analysis — Surgical video-documentation including continous iOCT will ne reviewed for Instrument tissue interactions at the grasp site of the starting point of Membrane peeling

SUMMARY:
Epiretinal membranes are a disease of the retinal surface, that may affect visual acuity and cause metamorphopsia. Using vitrectomy with membrane peeling, postoperative improvement of visual acuity and metamorphopsia may be achieved in a majority of patients. Diaz et al. demonstrated that there are postoperative changes in the "nerve fiber layer" after ILM peeling, but in that study, no recording of instrument/tissue interactions was performed using iOCT.

The aim of this study is to examine dipping into retinal tissue with the forceps during grasping of the epiretinal membrane at the starting point of peeling with iOCT.

DETAILED DESCRIPTION:
Epiretinal membranes are a disease of the retinal surface, that may affect visual acuity and cause metamorphopsia, occurring in approximately 20% of the population older than 60 years, as reported by Mitchell et al.. Using vitrectomy with membrane peeling, postoperative improvement of visual acuity and metamorphopsia may be achieved in a majority of patients. The surgical method has been used for some time, the first report on the surgical method of vitrectomy with membrane peeling was published by Machemer and dates back to 1978. Since the introduction of intraoperative optical coherence tomography (iOCT), intraoperative iatrogenically induced changes in retinal tissue can be detected and correlated with postoperative changes. Leisser et al. has been able to record "stretching" of the retinal tissue using this technique and has also been able to record the rarely occurring subfoveal and extrafoveal elevations of the ellipsoidal zone due to membrane peeling. These changes did not significantly affect postoperative visual acuity, according to Leisser et al., but did affect the development of postoperative microscotomas. Nevertheless, iOCT has the potential to document instrument tissue interactions such as dipping into retinal tissue with the forceps during grasping of the ERM at the starting point of membrane peeling. Diaz et al. demonstrated that there are postoperative changes in the "nerve fiber layer" after ILM peeling, but in that study, no recording of instrument/tissue interactions was performed using iOCT.

The aim of this study is to examine dipping into retinal tissue with the forceps during grasping of the epiretinal membrane at the starting point of peeling with iOCT.

ELIGIBILITY:
Inclusion Criteria:

* Vitrectomy with membrane peeling with iOCT assistance due to an ERM in the time-period from 1.6.2014 to 31.12.2016 (early phase) or 1.11.2020 to 31.7.2022.
* Age 18 and older

Exclusion Criteria:

* iOCT was not used during surgery
* bad image quality, excluding analysis of images

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical records of patients having undergone pars plana vitrectomy with Membrane Peeling and surgery assisted with iOCT in the time periods from 1.6.2014 to 31.12.2016 (early phase) or 1.11.2020 to 31.7.2022 (later phase) have been selected for data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
occurrence of dipping into retinal tissue with the ILM forceps during grasping | during surgery, an average of 30 minutes
  occurrence of dipping into retinal tissue during grasping will be evaluated (yes/no)
amount of dipping into retinal tissue with the ILM forceps during grasping, measured with ImageJ | during surgery, an average of 30 minutes
  amount of dipping into retinal tissue will be measured with calipers in ImageJ

SECONDARY OUTCOMES:
anatomical changes at the grasp site measured with optical coherence tomography | 3 months
  anatomical changes in retinal layers at the grasp site will be examinded by optical coherence tomography (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Leisser, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell P, Smith W, Chey T, Wang JJ, Chang A. Prevalence and associations of epiretinal membranes. The Blue Mountains Eye Study, Australia. Ophthalmology. 1997 Jun;104(6):1033-40. doi: 10.1016/s0161-6420(97)30190-0. PMID 9186446
- [Background] Machemer R. [The surgical removal of epiretinal macular membranes (macular puckers) (author's transl)]. Klin Monbl Augenheilkd. 1978 Jul;173(1):36-42. German. PMID 692034
- [Background] Leisser C, Palkovits S, Hienert J, Ullrich M, Zwickl H, Georgiev S, Findl O. Effect of Iatrogenic Traction during Macular Peeling Surgery on Postoperative Microperimetry. Ophthalmic Res. 2021;64(2):273-279. doi: 10.1159/000507633. Epub 2020 Apr 1. PMID 32235121
- [Background] Leisser C, Hackl C, Hirnschall N, Findl O. Effect of Subfoveal and Extrafoveal Hyporeflective Zones due to Iatrogenic Traction during Membrane Peeling for Epiretinal Membranes on Postoperative Outcomes. Ophthalmologica. 2020;243(4):297-302. doi: 10.1159/000505214. Epub 2019 Dec 5. PMID 31801147
- [Background] Diaz RI, Randolph JC, Sigler EJ, Calzada JI. Intraoperative grasp site correlation with morphologic changes in retinal nerve fiber layer after internal limiting membrane peeling. Ophthalmic Surg Lasers Imaging Retina. 2014 Jan-Feb;45(1):45-9. doi: 10.3928/23258160-20131220-06. PMID 24392911